CLINICAL TRIAL: NCT00626197
Title: A Randomised, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Two Doses of Ocrelizumab in Patients With WHO or ISN Class III or IV Nephritis Due to Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate Ocrelizumab in Patients With Nephritis Due to Systemic Lupus Erythematosus (BELONG)
Acronym: BELONG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to an imbalance of serious and opportunistic infections in the ocrelizumab treated patients versus the placebo arm.
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT4072g; WA20500
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Lupus Nephritis; Systemic Lupus Erythematosus
Keywords: SLE; Lupus; BELONG
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — Adrenal Cortex Hormones; Cyclophosphamide; Mycophenolic Acid; ocrelizumab; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- OCR 400 mg + SOC (Experimental): Participants received Ocrelizumab 400 mg i.v. infusion on Days 1 and 15, followed by 400 mg i.v. at Week 16 and then every 16 weeks plus SOC regimen.
  Interventions: Drug: Corticosteroids; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Ocrelizumab; Drug: Azathioprine
- OCR 1000 mg + SOC (Experimental): Participants received Ocrelizumab 1000 mg i.v. infusion on Days 1 and 15, followed by 1000 mg i.v. at Week 16 and then every 16 weeks plus SOC regimen.
  Interventions: Drug: Corticosteroids; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Ocrelizumab; Drug: Azathioprine
- Placebo + SOC (Placebo Comparator): Participants received placebo i.v. infusion on Days 1 and 15, followed by placebo infusion at Week 16 and then every 16 weeks plus SOC regimen.
  Interventions: Drug: Corticosteroids; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Placebo; Drug: Azathioprine

INTERVENTIONS:
Drug: Corticosteroids — Intravenous and oral repeating dose
Drug: Cyclophosphamide — Cyclophosphamide was administered at a IV dose 500 mg every 2 weeks for up to 6 doses followed by maintenance treatment with azathioprine.
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil was administered orally at maximum dose of 3 g/day.
Drug: Ocrelizumab — Ocrelizumab was administed at a dose and as per schedule in arm description
  Arms: OCR 1000 mg + SOC; OCR 400 mg + SOC
Drug: Placebo — Placebo was administered as per schedule in arm description
  Arms: Placebo + SOC
Drug: Azathioprine — Azathioprine was administered at a dose up to 2 mg/kg/day with a maximum dose of 200 mg.

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled, multicentre, parallel-group study designed to evaluate the efficacy and safety of ocrelizumab added to SOC (corticosteroid plus one of two immunosuppressant regimens) compared with placebo added to SOC in patients with WHO or ISN Class III or IV lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or above at the time of the screening
* Ability and willingness to provide written informed consent and to comply with the schedule of protocol requirements
* Diagnosis of SLE
* Active lupus nephritis

Exclusion Criteria:

* Currently active retinitis, poorly controlled seizure disorder, acute confusional state, myelitis, stroke or stroke syndrome, cerebellar ataxia, or dementia
* Severe renal impairment
* Lack of peripheral venous access
* Pregnancy or breast feeding mothers
* History of severe allergic or anaphylactic reactions to humanized, chimeric or murine monoclonal antibodies or i.v. immunoglobulin
* Known severe chronic pulmonary disease
* Evidence of significant uncontrolled concomitant diseases in any organ system not related to SLE, which, in the investigator's opinion, would preclude patient participation
* Concomitant condition which has required treatment with systemic corticosteroid (excluding topical or inhaled steroids) prior to screening
* Known HIV or chronic active Hepatitis B or chronic active Hepatitis C infection
* Known active infection of any kind prior to Day 1
* History of serious recurrent or chronic infection
* History of cancer, including solid tumors, hematological malignancies and carcinoma in situ (except basal cell carcinoma of the skin that has been excised and cured).
* History of alcohol or drug abuse prior to screening
* Major surgery prior to screening, excluding diagnostic surgery
* Previous treatment with CAMPATH-1H
* Previous treatment with a BAFF directed treatment (e.g. anti-BLyS) prior to screening
* Previous treatment with a B-cell targeted therapy other than one directed at BAFF (e.g. anti-CD20, anti-CD22)
* Treatment with any investigational agent prior to screening
* Receipt of any live vaccines prior to Day 1
* Intolerance or contraindication to oral or i.v. corticosteroids
* Positive hepatitis BsAg or hepatitis C serology. Patients who are HBsAg negative but HBcAb positive may be enrolled with a negative DNA test

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2008-02-15 (Actual); Primary Completion 2009-10-19 (Actual); Study Completion 2013-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening was done from Day -14 to Day -1.
Groups:
- OCR 400 mg + SOC: Participants received 400 mg ocrelizumab IV on Days 1 and 15, followed by 400 mg ocrelizumab infusion IV on Week 16 and then every 16 weeks up to 48 weeks along with one of the two standard-of-care (SOC) immunosuppressant regimens at the discretion of the investigator. The SOC regimens were: Euro-Lupus (cyclophosphamide 500 mg every 2 weeks for 6 doses followed by azathioprine maintenance at 1-2 milligrams per kilogram per day [mg/kg/day]), or MMF 1 g/day in the first week increased to 3 g/day. Participants also received methylprednisolone 100 mg infusion IV or according to local guidelines, completed at least 30 minutes prior to each infusion of ocrelizumab. Participants also received oral prednisone at starting dose of 0.75 mg/kg/day with a maximum dose of 60 mg/day from Day 2. Beginning on Day 16 the doses were tapered and continued for 10 weeks to a target dose of 10 mg/day.
- OCR 1000 mg + SOC: Participants received 1000 mg ocrelizumab IV on Days 1 and 15, followed by 1000 mg ocrelizumab infusion IV on Week 16 and then every 16 weeks up to 48 weeks along with one of the two standard-of-care (SOC) immunosuppressant regimens at the discretion of the investigator. The SOC regimens were: Euro-Lupus (cyclophosphamide 500 mg every 2 weeks for 6 doses followed by azathioprine maintenance at 1-2 milligrams per kilogram per day [mg/kg/day]), or MMF 1 g/day in the first week increased to 3 g/day. Participants also received methylprednisolone 100 mg infusion IV or according to local guidelines, completed at least 30 minutes prior to each infusion of ocrelizumab. Participants also received oral prednisone at starting dose of 0.75 mg/kg/day with a maximum dose of 60 mg/day from Day 2. Beginning on Day 16 the doses were tapered and continued for 10 weeks to a target dose of 10 mg/day.
- Placebo + SOC: Participants received placebo matched to ocrelizumab infusion intravenously (IV) on Days 1 and 15, followed by placebo matched to ocrelizumab infusion IV on Week 16 and then every 16 weeks up to 48 weeks along with one of the two standard-of-care (SOC) immunosuppressant regimens at the discretion of the investigator. The SOC regimens were: Euro-Lupus (cyclophosphamide 500 mg every 2 weeks for 6 doses followed by azathioprine maintenance at 1-2 milligrams per kilogram per day [mg/kg/day]), or mycophenolate mofetil (MMF) 1 grams per day (g/day) in the first week increased to 3 g/day. Participants also received methylprednisolone 100 milligram (mg) infusion IV or according to local guidelines, completed at least 30 minutes prior to each infusion of placebo. Participants also received oral prednisone at a starting dose of 0.75 mg/kg/day with a maximum dose of 60 mg/day from Day 2. Beginning on Day 16 the doses were tapered and continued for 10 weeks to a target dose of 10 mg/day.
Period: Overall Study
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Started | 127 | 128 | 126
Completed | 83 | 74 | 49
Not Completed | 44 | 54 | 77
Not completed — Did not cooperate | 2 | 6 | 1
Not completed — Failure to return | 6 | 5 | 6
Not completed — Adverse event, serious fatal | 3 | 6 | 6
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Withdrawal by Subject | 17 | 17 | 7
Not completed — Administrative reasons | 15 | 19 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 127 | 128 | 126 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.9 (10.2) | 30.6 (8.9) | 31.3 (9.9) | 31.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 110 | 107 | 332
  Male | 12 | 18 | 19 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 15 | 17 | 49
  Asian | 39 | 27 | 35 | 101
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 5 | 19
  White | 55 | 67 | 58 | 180
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 12 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Complete Renal Response (CRR)
Description: CRR was defined as: 1. Normal serum creatinine (and with no more than a 25 percent [%] increase from Baseline); 2. Improvement in urinary protein:urinary creatinine ratio to less than or equal to (≤) 0.5. PRR was defined as at least 50 percent (%) reduction in proteinuria from Baseline, without more than 25% increase of serum creatinine at Week 48, compared with Baseline. If Baseline urine protein:urine creatinine ratio was greater than (>) 3, a urine protein:urine creatinine ratio of less than (<) 3 needed to be achieved.
Time Frame: Week 48
Population: The primary endpoint was analyzed via an overall response (CRR+PRR) analysis and the separate complete and partial response rates were only summarized descriptively
Measure: Number; unit: Percentage of Participants
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 75 | 73 | 75
Percentage of Participants
  CRR | 42.7 | 31.5 | 34.7
  PRR | 24 | 35.6 | 20

2. Primary Outcome: Percentage of Participants Who Achieved Overall Response
Description: Overall response rate (ORR) equals (=) CRR + PRR. CRR was defined as: 1. Normal serum creatinine (and with no more than a 25% increase from baseline) 2. Improvement in urinary protein:urinary creatinine ratio to ≤0.5. PRR was defined as at least 50 % reduction in proteinuria from Baseline, without more than 25% increase of serum creatinine at Week 48, compared with Baseline. If Baseline urine protein:urine creatinine ratio is >3, a urine protein:urine creatinine ratio of <3 needs to be achieved.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 75 | 73 | 75
Percentage of Participants | 66.7 [56 to 77.3] | 67.1 [56.3 to 77.9] | 54.7 [43.4 to 65.9]

3. Secondary Outcome: Percentage of Participants Who Achieved a Renal Response (Partial or Complete) by Week 36, and Sustain or Improve This Response Until Week 48
Time Frame: Weeks 36, 40, 44, and 48
Population: Efficacy date were summarized in the primary endpoints and due to early study termination the protocol was modified to transition the participants into the safety follow-up period. Additional efficacy outcome measures were not analyzed and study results focus on the full summary of safety data.
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time To Complete Renal Response
Description: Time to complete renal response was proposed to be analyzed using a stratified log rank test with race and SOC as stratification factors. Comparisons of ocrelizumab versus placebo were to be expressed as p-values, estimated hazard ratios, adjusted proportions of participants who achieved a complete renal response and their 95% confidence intervals. Kaplan-Meier curves were to be produced. Due to early termination of the study the analyses were not performed.
Time Frame: Baseline up to Week 48
Population: as for outcome 3
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Area Under the Curve (AUC) of Calculated Glomerular Filtration Rate (cGFR) Between Baseline and Week 48
Description: The improvement of AUC of cGFR was to be measured between Baseline and Week 48. This was to be analyzed with Analysis of Covariance (ANCOVA) with race and SOC as covariates.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and Week 48
Population: Due to the early termination and unblinding of the study, no data was collected for this endpoint and analysis was not performed.
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Achieved A Reduction In Systemic Lupus Erythematosis Disease Activity Index (SLEDAI) -2K Score
Description: SLEDAI-2K measures disease activity at the visit or within the preceding 10 days. It comprised of 24 descriptors, covering 9 organ systems, and reflects disease activity over the previous 10 days.The total SLEDAI-2K score falls between 0 and 105, with higher scores representing higher disease activity
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Time to First Renal Flare In Those Participants Who Demonstrated at Least a Partial Renal Response
Description: Renal flares may be either proteinuric or nephritic as defined below: Proteinuric Flares are defined as follows:In participants who achieve a urine protein:urine creatinine (Upr:Ucr) ≤ 0.5, an increase to Upr:Ucr >1; In participants with an Upr:Ucr >0.5, a doubling of Upr:Ucr (with a minimum increase to Upr:Ucr >2). Nephritic Flare defined as: Increase in serum creatinine of ≥30% from the lowest value achieved in the study accompanied by Increase Upr:Ucr >1 Or New/worsening active urine sediment on two consecutive occasions, in the absence of urinary tract infection or other causes of hematuria.
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 3
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Who Achieved Clinically Meaningful Improvement in the Physical and Mental Component Scores of the Short Form 36 (SF36) From Baseline to Week 48
Description: The SF36 Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions physical role functioning, emotional role functioning, social role functioning, and mental health.
Time Frame: Baseline and Weeks 1, 12, 24, 36, and 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants Who Achieved Clinically Meaningful Improvement in Fatigue Using the Functional Assessment of Chronic Illness Therapy (Facit) Fatigue Questionnaire From Baseline to Week 48
Description: The FACIT Fatigue Scale is a short, 13-item, easy-to-administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued).
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants Who Achieved Clinically Meaningful Improvement in Pain Using the Modified Brief Pain Inventory Short Form (mBPI-SF) From Baseline to Week 48
Description: m-BPI-sf is a self-administered 11-point Likert rating scale to rate pain in the past 24 hours. A single item pertains to worst pain in the past 24 hours with a range of 0 (no pain) to 10 (worst imaginable pain).
Time Frame: Baseline and Weeks 1, 12, 24, 36, and 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Health Care Visits Over the 48-Week Treatment Period
Description: The number of health care visits (including doctor's office visits, Emergency room/ Accident and Emergency [ER/A&E] visits and hospitalizations) over the 48-week treatment period were recorded.
Time Frame: Weeks 1, 24, and 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants Who Achieved a CRR or PRR And Who Received A Corticosteroid Dose of <10 Milligrams Per Day (mg/Day) From Week 24 to Week 48
Description: CRR was defined as: 1. Normal serum creatinine (and with no more than a 25% increase from Baseline) 2. Inactive urinary sediment 3. Improvement in urinary protein:urinary creatinine ratio to ≤0.5. PRR was defined as at least 50% reduction in proteinuria from Baseline, without more than 25% increase of serum creatinine at Week 48, compared with Baseline. If Baseline urine protein:urine creatinine ratio was >3, a urine protein:urine creatinine ratio of <3 needed to be achieved.
Time Frame: Week 48
Population: as for outcome 3
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants Who Achieved a CRR or PRR And Who Received a Corticosteroid Dose of <5 mg/Day by Week 48
Description: CRR was defined as: 1. Normal serum creatinine (and with no more than a 25% increase from Baseline) 2. Inactive urinary sediment 3. Improvement in urinary protein:urinary creatinine ratio to ≤0.5. PRR was defined as at least 50% reduction in proteinuria from Baseline, without more than 25% increase of serum creatinine at Week 48, compared with Baseline. If Baseline urine protein:urine creatinine ratio was >3, a urine protein: urine creatinine ratio of <3 needed to be achieved.
Time Frame: Week 48
Population: as for outcome 3
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Average Corticosteroid Burden Measured by AUC of the Cumulative Corticosteroid Dose Between 16 and 48 Weeks
Description: AUC is the area under the curve (mathematically known as definite integral) in a plot of concentration of drug in blood plasma against time. AUC was to be used to determine the average corticosteroid burden.
Time Frame: Weeks 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants Who Stopped Immunosuppressants After Week 48
Description: The number of participants who stopped immunosuppressants were to be determined by survey.
Time Frame: Week 48
Population: as for outcome 5
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Mean Absolute Counts of Cluster of Differentiation (CD) 19 Positive (+) Cells Per Visit
Description: CD19 is a cell surface molecule which assembles with the antigen receptor of B lymphocytes. It is a critical signal transduction molecule that regulates B lymphocyte development, activation, and differentiation. CD19+ cells were measured as cells per microliter (cells/uL).
Time Frame: Baseline, Day 15, Week 4, 16, 32, 48, and by infusion (pre and post infusion) on Day 1, 15, Week 16, 32
Population: N = number of participants analyzed at the specified visit
Measure: Mean (Standard Deviation); unit: Cells/uL
Groups:
- OCR + SOC: This analysis set included all participants who were treated with ocrelizumab (OCR).
- Placebo-Mycophenolate Mofetil (MMF): Placebo - MMF group included participants whose SOC treatment included MMF as an immunosuppressant treatment.
- Placebo-Euro Lupus (EL): Placebo-EL group included participants whose SOC treatment included Cyclophosphamide (Euro-lupus) as part of the immunosuppressant treatment.
Arm/Group | Placebo + SOC | OCR 400 mg + SOC | OCR 1000 mg + SOC | OCR + SOC | Placebo-Mycophenolate Mofetil (MMF) | Placebo-Euro Lupus (EL)
Number analyzed (Participants) | 75 | 73 | 70 | 141 | 45 | 27
Cells/uL
  Baseline: number analyzed (Participants) | 75 | 71 | 66 | 137 | 44 | 26
  Baseline | 203.5 (191.4) | 256.3 (300.2) | 224.1 (231.7) | 240.8 (268.9) | 213.7 (201.7) | 186.3 (175)
  Day 15: number analyzed (Participants) | 66 | 70 | 68 | 138 | 40 | 26
  Day 15 | 262.7 (273.9) | 1.9 (1.9) | 2.2 (3.4) | 2 (2.7) | 327.4 (324.9) | 163.3 (115.8)
  Week 4: number analyzed (Participants) | 68 | 67 | 67 | 134 | 41 | 27
  Week 4 | 209.7 (221.4) | 1.4 (2.5) | 1.3 (1.6) | 1.4 (2.1) | 253.4 (263.9) | 143.3 (107.4)
  Week 16: number analyzed (Participants) | 70 | 72 | 69 | 141 | 45 | 25
  Week 16 | 125.9 (186.9) | 2.6 (3.6) | 2 (3.8) | 2.3 (3.7) | 154.3 (222.2) | 74.7 (75.3)
  Week 32: number analyzed (Participants) | 68 | 73 | 68 | 141 | 45 | 23
  Week 32 | 116.6 (154.3) | 7.8 (25.8) | 2.1 (2.7) | 5.1 (18.8) | 141.2 (172.5) | 68.5 (96.8)
  Week 48: number analyzed (Participants) | 68 | 71 | 66 | 137 | 45 | 23
  Week 48 | 110 (114.3) | 11.7 (43.6) | 2.6 (8.9) | 7.3 (32.2) | 134.9 (123.3) | 61.3 (75)
  Day 1 Pre-infusion: number analyzed (Participants) | 75 | 71 | 67 | 138 | 44 | 26
  Day 1 Pre-infusion | 203.5 (191.4) | 256.3 (300.2) | 222.8 (230.2) | 240 (268) | 213.7 (201.7) | 186.3 (175)
  Day 1 Post-infusion: number analyzed (Participants) | 70 | 69 | 68 | 137 | 43 | 27
  Day 1 Post-infusion | 103.1 (115.1) | 11.1 (28.6) | 5.7 (8.5) | 8.4 (21.3) | 102.4 (114.3) | 104.3 (118.6)
  Day 15 Pre-infusion: number analyzed (Participants) | 68 | 68 | 70 | 138 | 43 | 25
  Day 15 Pre-infusion | 264.4 (276.6) | 1.9 (1.9) | 2.1 (3.3) | 2 (2.7) | 322.5 (323.5) | 164.5 (118)
  Day 15 Post-infusion: number analyzed (Participants) | 67 | 65 | 68 | 133 | 42 | 25
  Day 15 Post-infusion | 91.2 (109.2) | 1 (1.3) | 0.9 (1.4) | 0.9 (1.3) | 106.3 (130.8) | 65.8 (50.4)
  Week 16 Pre-infusion: number analyzed (Participants) | 67 | 66 | 66 | 132 | 43 | 24
  Week 16 Pre-infusion | 127.8 (190.1) | 2.5 (3.3) | 2.1 (3.9) | 2.3 (3.6) | 156.5 (226.3) | 76.3 (76.5)
  Week 16 Post-infusion: number analyzed (Participants) | 61 | 66 | 66 | 132 | 40 | 21
  Week 16 Post-infusion | 52.7 (72.6) | 1.2 (1.6) | 0.8 (1) | 1 (1.3) | 64.2 (83) | 30.9 (40.2)
  Week 32 Pre-infusion: number analyzed (Participants) | 60 | 63 | 63 | 126 | 39 | 21
  Week 32 Pre-infusion | 125 (161.1) | 5.1 (16.5) | 2 (2.7) | 3.6 (11.8) | 153.4 (180.6) | 72.2 (100.4)
  Week 32 Post-infusion: number analyzed (Participants) | 60 | 63 | 59 | 122 | 38 | 22
  Week 32 Post-infusion | 46.2 (54.4) | 1 (1.5) | 0.7 (1.4) | 0.9 (1.4) | 56.9 (62.5) | 27.6 (29.5)

17. Secondary Outcome: Percentage of Participants With CD19+ Absolute B Cell Counts <10 Cells Per Microliter (Cells/uL)
Description: CD19 is a cell surface molecule which assembles with the antigen receptor of B lymphocytes. It is a critical signal transduction molecule that regulates B lymphocyte development, activation, and differentiation. 0 represents 0% of participants.
Time Frame: Baseline, Day 15, Week 4, 16, 32, 48, and by infusion (pre and post infusion) on Day 1, 15, Week 16, 32
Population: N = number of participants analyzed at the specified visit
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + SOC | OCR 400 mg + SOC | OCR 1000 mg + SOC | OCR + SOC | Placebo-Mycophenolate Mofetil (MMF) | Placebo-Euro Lupus (EL)
Number analyzed (Participants) | 75 | 75 | 73 | 148 | 47 | 28
Percentage of Participants
  Baseline: number analyzed (Participants) | 75 | 71 | 66 | 137 | 44 | 26
  Baseline | 4.3 | 4.2 | 1.5 | 2.9 | 6.8 | 0
  Day 15: number analyzed (Participants) | 66 | 70 | 68 | 138 | 40 | 26
  Day 15 | 4.5 | 100 | 97.1 | 98.6 | 7.5 | 0
  Week 4: number analyzed (Participants) | 68 | 67 | 67 | 134 | 41 | 27
  Week 4 | 4.4 | 98.5 | 100 | 99.3 | 7.3 | 0
  Week 16: number analyzed (Participants) | 70 | 72 | 69 | 141 | 45 | 25
  Week 16 | 4.3 | 95.8 | 97.1 | 96.5 | 6.7 | 0
  Week 32: number analyzed (Participants) | 68 | 73 | 68 | 141 | 45 | 23
  Week 32 | 7.4 | 91.8 | 95.6 | 93.6 | 8.9 | 4.3
  Week 48: number analyzed (Participants) | 68 | 71 | 66 | 137 | 45 | 23
  Week 48 | 5.9 | 88.7 | 98.5 | 93.4 | 4.4 | 8.7
  Day 1 Pre-infusion: number analyzed (Participants) | 75 | 71 | 67 | 138 | 44 | 26
  Day 1 Pre-infusion | 4.3 | 4.2 | 1.5 | 2.9 | 6.8 | 0
  Day 1 Post-infusion: number analyzed (Participants) | 70 | 69 | 68 | 137 | 43 | 28
  Day 1 Post-infusion | 10 | 81.2 | 83.8 | 82.5 | 14 | 3.7
  Day 15 Pre-infusion: number analyzed (Participants) | 68 | 68 | 70 | 138 | 43 | 25
  Day 15 Pre-infusion | 4.4 | 100 | 97.1 | 98.6 | 7 | 0
  Day 15 Post-infusion: number analyzed (Participants) | 67 | 65 | 68 | 133 | 42 | 25
  Day 15 Post-infusion | 7.5 | 100 | 100 | 100 | 11.9 | 0
  Week 16 Pre-infusion: number analyzed (Participants) | 67 | 66 | 66 | 132 | 43 | 24
  Week 16 Pre-infusion | 4.5 | 97 | 97 | 97 | 7 | 0
  Week 16 Post-infusion: number analyzed (Participants) | 61 | 66 | 66 | 132 | 40 | 21
  Week 16 Post-infusion | 11.5 | 100 | 100 | 100 | 12.5 | 9.5
  Week 32 Pre-infusion: number analyzed (Participants) | 60 | 63 | 63 | 126 | 39 | 21
  Week 32 Pre-infusion | 3.3 | 93.7 | 95.2 | 94.4 | 5.1 | 0
  Week 32 Post-infusion: number analyzed (Participants) | 60 | 63 | 59 | 122 | 38 | 22
  Week 32 Post-infusion | 15 | 100 | 100 | 100 | 10.5 | 22.7

18. Secondary Outcome: Percentage of Participants With CD19+ Absolute B Cell Counts <20 Cells/uL by Visit
Description: CD19 is a cell surface molecule which assembles with the antigen receptor of B lymphocytes. It is a critical signal transduction molecule that regulates B lymphocyte development, activation, and differentiation. n = number of participants analyzed at the specified visit. 0 represents 0% of participants.
Time Frame: Baseline, Day 15, Week 4, 16, 32, 48, and by infusion (pre and post infusion) on Day 1, 15, Week 16, 32
Population: N = number of participants analyzed at the specified visit
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + SOC | OCR 400 mg + SOC | OCR 1000 mg + SOC | OCR + SOC | Placebo-Mycophenolate Mofetil (MMF) | Placebo-Euro Lupus (EL)
Number analyzed (Participants) | 75 | 75 | 73 | 148 | 47 | 28
Percentage of Participants
  Baseline: number analyzed (Participants) | 70 | 71 | 66 | 137 | 44 | 26
  Baseline | 7.1 | 11.3 | 3 | 7.3 | 11.4 | 0
  Day 15: number analyzed (Participants) | 66 | 70 | 68 | 138 | 40 | 26
  Day 15 | 7.6 | 100 | 98.5 | 99.3 | 10 | 3.8
  Week 4: number analyzed (Participants) | 68 | 67 | 67 | 134 | 41 | 27
  Week 4 | 10.3 | 100 | 100 | 100 | 12.2 | 7.4
  Week 16: number analyzed (Participants) | 70 | 72 | 69 | 141 | 45 | 25
  Week 16 | 11.4 | 98.6 | 98.6 | 98.6 | 13.3 | 8
  Week 32: number analyzed (Participants) | 68 | 73 | 68 | 141 | 45 | 23
  Week 32 | 13.2 | 93.2 | 100 | 96.5 | 15.6 | 8.7
  Week 48: number analyzed (Participants) | 68 | 71 | 66 | 137 | 45 | 23
  Week 48 | 17.6 | 91.5 | 98.5 | 94.9 | 13.3 | 26.1
  Day 1 Pre-infusion: number analyzed (Participants) | 75 | 71 | 67 | 138 | 44 | 26
  Day 1 Pre-infusion | 7.1 | 11.3 | 3 | 7.2 | 11.4 | 0
  Day 1 Post-infusion: number analyzed (Participants) | 70 | 69 | 68 | 137 | 43 | 28
  Day 1 Post-infusion | 22.9 | 87 | 91.2 | 89.1 | 20.9 | 25.9
  Day 15 Pre-infusion: number analyzed (Participants) | 68 | 68 | 70 | 138 | 43 | 25
  Day 15 Pre-infusion | 7.4 | 100 | 98.6 | 99.3 | 9.3 | 4
  Day 15 Post-infusion: number analyzed (Participants) | 67 | 65 | 68 | 133 | 42 | 25
  Day 15 Post-infusion | 17.9 | 100 | 100 | 100 | 21.4 | 12
  Week 16 Pre-infusion: number analyzed (Participants) | 67 | 66 | 66 | 132 | 43 | 24
  Week 16 Pre-infusion | 10.4 | 98.5 | 98.5 | 98.5 | 11.6 | 8.3
  Week 16 Post-infusion: number analyzed (Participants) | 61 | 66 | 66 | 132 | 40 | 21
  Week 16 Post-infusion | 41 | 100 | 100 | 100 | 32.5 | 57.1
  Week 32 Pre-infusion: number analyzed (Participants) | 60 | 63 | 63 | 126 | 39 | 21
  Week 32 Pre-infusion | 8.3 | 95.2 | 100 | 97.6 | 10.3 | 4.8
  Week 32 Post-infusion: number analyzed (Participants) | 60 | 63 | 59 | 122 | 38 | 22
  Week 32 Post-infusion | 35 | 100 | 100 | 100 | 26.3 | 50

19. Secondary Outcome: Percentage of Participants With CD19+ Absolute B Cell Counts Less Than the Lower Limit of Normal (LLN) by Visit
Description: CD19 is a cell surface molecule which assembles with the antigen receptor of B lymphocytes. It is a critical signal transduction molecule that regulates B lymphocyte development, activation, and differentiation. <LLN = 80 cells/uL.
Time Frame: Baseline, Day 15, Week 4, 16, 32, 48, and by infusion (pre and post infusion) on Day 1, 15, Week 16, 32
Population: N = number of participants analyzed at the specified visit
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + SOC | OCR 400 mg + SOC | OCR 1000 mg + SOC | OCR + SOC | Placebo-Mycophenolate Mofetil (MMF) | Placebo-Euro Lupus (EL)
Number analyzed (Participants) | 70 | 73 | 70 | 141 | 45 | 27
Percentage of Participants
  Baseline: number analyzed (Participants) | 70 | 71 | 66 | 137 | 44 | 26
  Baseline | 27.1 | 36.6 | 33.3 | 35 | 29.5 | 23.1
  Day 15: number analyzed (Participants) | 66 | 70 | 68 | 138 | 40 | 26
  Day 15 | 28.8 | 100 | 100 | 100 | 30 | 26.9
  Week 4: number analyzed (Participants) | 68 | 67 | 67 | 134 | 41 | 27
  Week 4 | 39.7 | 100 | 100 | 100 | 39 | 40.7
  Week 16: number analyzed (Participants) | 70 | 72 | 69 | 141 | 45 | 25
  Week 16 | 57.1 | 100 | 100 | 100 | 48.9 | 72
  Week 32: number analyzed (Participants) | 68 | 73 | 68 | 141 | 45 | 23
  Week 32 | 52.9 | 97.3 | 100 | 98.6 | 35.6 | 87
  Week 48: number analyzed (Participants) | 68 | 71 | 66 | 137 | 45 | 23
  Week 48 | 51.5 | 97.2 | 100 | 98.5 | 37.8 | 78.3
  Day 1 Pre-infusion: number analyzed (Participants) | 70 | 71 | 67 | 138 | 44 | 26
  Day 1 Pre-infusion | 27.1 | 36.6 | 32.8 | 34.8 | 29.5 | 23.1
  Day 1 Post-infusion: number analyzed (Participants) | 70 | 69 | 68 | 137 | 43 | 27
  Day 1 Post-infusion | 55.7 | 97.1 | 100 | 98.5 | .5 | 59.3
  Day 15 Pre-infusion: number analyzed (Participants) | 68 | 68 | 70 | 138 | 43 | 25
  Day 15 Pre-infusion | 30.0 | 100 | 100 | 100 | 32.6 | 28
  Day 15 Post-infusion: number analyzed (Participants) | 67 | 65 | 68 | 133 | 42 | 25
  Day 15 Post-infusion | 58.2 | 100 | 100 | 100 | 52.4 | 68
  Week 16 Pre-infusion: number analyzed (Participants) | 67 | 66 | 66 | 132 | 43 | 24
  Week 16 Pre-infusion | 56.7 | 100 | 100 | 100 | 48.8 | 70.8
  Week 16 Post-infusion: number analyzed (Participants) | 61 | 66 | 66 | 132 | 40 | 21
  Week 16 Post-infusion | 80.3 | 100 | 100 | 100 | 72.5 | 95.2
  Week 32 Pre-infusion: number analyzed (Participants) | 60 | 63 | 63 | 126 | 39 | 21
  Week 32 Pre-infusion | 50 | 98.4 | 100 | 99.2 | 30.8 | 85.7
  Week 32 Post-infusion: number analyzed (Participants) | 60 | 63 | 59 | 122 | 38 | 22
  Week 32 Post-infusion | 88.3 | 100 | 100 | 100 | 84.2 | 95.5

20. Secondary Outcome: Percentage of Participants Achieving a Major Clinical Response or a Partial Clinical Response
Description: A major clinical response was defined as British Isles Lupus Assessment Group (BILAG) C scores or better at Week 24 without developing any new A or two new B scores up to Week 24 and maintenance of this response without developing a moderate or severe flare between Week 24 and Week 48. A partial clinical response was defined as BILAG C scores or better at Week 24 and maintaining this response without developing a flare for 16 consecutive weeks. The BILAG is an organ-specific 86-question assessment based on the principle of the doctor's intent to treat, which requires an assessment of improved (1), the same (2), worse (3), or new (4) over the last month. Within each organ system, multiple manifestations and laboratory tests are combined into a single score for that organ. The resulting scores for each organ can be A through E, where A is very active disease, B is moderate activity, C is mild stable disease, D is resolved activity, and E indicates the organ was never involved.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 3
Arm/Group | OCR 400 mg + SOC | OCR 1000 mg + SOC | Placebo + SOC
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 19 months.
Description: All patients who received any part of an infusion of study drug and provided at least one assessment of safety were included in the safety analysis.
Arm/Group | Placebo + SOC | OCR 1000 mg + SOC | OCR 400 mg + SOC
All-Cause Mortality (participants affected / at risk) | 6/125 | 6/127 | 3/126
Serious Adverse Events (participants affected / at risk) | 36/125 | 38/127 | 53/126
Other Adverse Events (participants affected / at risk) | 96/125 | 91/127 | 101/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SOC (N=125) | OCR 1000 mg + SOC (N=127) | OCR 400 mg + SOC (N=126)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Polyserositis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lupus encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Vasculitis cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (2) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (5) | 3 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (3) | 5 (5)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (11)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Legionella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neurocryptococcosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 8 (8) | 4 (5)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Strongyloidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SOC (N=125) | OCR 1000 mg + SOC (N=127) | OCR 400 mg + SOC (N=126)
Hypertension (Vascular disorders) | 7 (8) | 12 (15) | 12 (19)
Infusion related reaction (Injury, poisoning and procedural complications) | 11 (12) | 17 (19) | 14 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5) | 11 (12)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 7 (7) | 13 (17)
Leukopenia (Blood and lymphatic system disorders) | 7 (11) | 12 (17) | 18 (24)
Neutropenia (Blood and lymphatic system disorders) | 6 (7) | 7 (10) | 15 (27)
Dizziness (Nervous system disorders) | 9 (9) | 5 (6) | 6 (6)
Headache (Nervous system disorders) | 11 (18) | 11 (12) | 15 (21)
Oedema peripheral (General disorders) | 8 (9) | 4 (4) | 2 (5)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 7 (7)
Insomnia (Psychiatric disorders) | 3 (4) | 7 (7) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 7 (8) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 22 (29) | 32 (36) | 26 (35)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 3 (3) | 9 (10)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (3) | 11 (15)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (5) | 13 (16)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (8) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) | 6 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 8 (8)
Dyslipidaemia (Metabolism and nutrition disorders) | 11 (14) | 2 (2) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (12) | 4 (4) | 9 (16)
Bronchitis (Infections and infestations) | 10 (16) | 10 (12) | 14 (17)
Gastroenteritis (Infections and infestations) | 10 (11) | 4 (4) | 7 (10)
Herpes zoster (Infections and infestations) | 6 (6) | 9 (11) | 8 (9)
Nasopharyngitis (Infections and infestations) | 16 (23) | 13 (20) | 17 (24)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 7 (10)
Pharyngitis (Infections and infestations) | 4 (4) | 7 (7) | 13 (13)
Sinusitis (Infections and infestations) | 3 (4) | 7 (12) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 19 (28) | 23 (43) | 22 (42)
Urinary tract infection (Infections and infestations) | 13 (13) | 18 (35) | 24 (43)

LIMITATIONS AND CAVEATS:
The study was terminated early due to an imbalance in serious infections in ocrelizumab-treated participants versus placebo-treated participants. Only 139 of the 381 participants randomized completed the 48 week treatment period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.